CLINICAL TRIAL: NCT02012140
Title: Pharmacokinetics and Pharmacodynamics of Ticagrelor in Patients With Stable Angina, NSTEMI and STEMI Undergoing PCI
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: LifeBridge Health (Other)
Responsible Party: Principal Investigator, Paul A. Gurbel, Director, LifeBridge Health
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AZSC01
Record Dates: First submitted 2013-11-05; First posted 2013-12-16 (Estimated); Last update posted 2013-12-16 (Estimated); Status verified 2013-12

CONDITIONS: Cardiovascular Disease; Stable Angina; Myocardial Infarction; Coronary Artery Disease
MeSH Terms: conditions — Cardiovascular Diseases; Angina, Stable; Myocardial Infarction; Coronary Artery Disease | interventions — Ticagrelor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ticagrelor (Experimental): As per ACC/AHA and ESC guidelines 180 mg is the recommended LD. The ticagrelor 90 mg BID dose, following the loading dose, has been selected for the clopidogrel naïve patients with stable angina, NSTEMI and STEMI patients undergoing PCI as the maintenance dose for this study since it is the FDA recommended dose.
  Interventions: Drug: ticagrelor

INTERVENTIONS:
Drug: ticagrelor

SUMMARY:
Ticagrelor therapy has been shown to reduce the rates of cardiovascular events and all-cause mortality compared to clopidogrel therapy in patients with acute coronary syndromes (ACS). The benefit of this study would be to demonstrate that ticagrelor therapy is associated with equivalent platelet inhibition irrespective of the disease status in patients undergoing PCI.

ELIGIBILITY:
Inclusion Criteria:

* Stable Angina: Stable coronary artery disease patients with documented ischemia undergoing elective PCI will be enrolled.Inclusion criteria for enrollment in the ACS group with or without ST-segment elevation, requires onset of symptoms during the previous 48 hours.

NSTEMI

For patients who had an ACS without ST-segment elevation (NTSEMI), two of the following criteria had to be met:

* a positive test of a biomarker (troponin I) in accordance with the universal definitions indicating myocardial necrosis
* ST-segment changes on electrocardiography, indicating ischemia that do not meet criteria for STEMI.

STEMI

For patients who had an ACS with ST-segment elevation, the following two inclusion criteria had to be met:

* either persistent ST-segment elevation of at least 0.1 mV in at least two contiguous leads or a new left bundle-branch block; and
* the intention to perform primary PCI with 24 hours of symptom onset

Exclusion Criteria:

* Patients who are on P2Y12 receptor blockers, oral anticoagulants, or GPIIb/IIIa receptor blocker therapies.
* Presence or history of any of the following: ischemic or hemorrhagic stroke; transient ischemic attack (TIA); intracranial neoplasm; arteriovenous malformation, or aneurysm; intracranial hemorrhage; head trauma (within 3 months of study entry)
* History of refractory ventricular arrhythmias or an increased risk of bradycardic events (eg, subjects without a pacemaker who have sick sinus syndrome, 2nd or 3rd degree atrioventricular (AV) block or bradycardic-related syncope)
* History or evidence of congestive heart failure (New York Heart Association Class III or above ≤ 6 months before screening
* Severe hepatic impairment defined as ALT> 2.5 X ULN
* Uncontrolled hypertension, or systolic blood pressure > 180 mmHg or diastolic blood pressure > 110 mmHg at screening
* Severely impaired renal function (glomerular filtration rate < 30 mL/minute) or on dialysis
* Platelet count <100 X103, illicit drug or alcohol abuse, prothrombin time>1.5 times control, haematocrit <30%, and creatinine >2.0 mg/dl.
* Contraindication or other reason that ticagrelor should not be administered (eg, hypersensitivity, active bleeding, moderate or severe liver disease, history of previous intracranial bleed, GI bleed within the past 6 months, major surgery within 30 days)
* Fibrinolytic therapy in the 24 hours prior to PCI, or planned fibrinolytic treatment following PCI.
* Participation in another investigational drug or device study in the last 30 -Pregnancy or lactation
* Concomitant oral or intravenous therapy (see examples below) with strong CYP3A inhibitors, CYP3A substrates with narrow therapeutic indices, or strong CYP3A inducers which cannot be stopped for the course of the study
* Strong inhibitors: ketoconazole, itraconazole, voriconazole, telithromycin, clarithromycin, nefazadone, ritonavir, saquinavir, nelfinavir, indinavir, atanazavir
* Substrates with narrow therapeutic index: cyclosporine, quinidine
* Strong inducers: rifampin/rifampicin, phenytoin, carbamazepine
* Any other condition which in the opinion of the investigator, may either put the patient at risk or influence the result of the study (eg, cardiogenic shock or severe haemodynamic instability, active cancer, risk for non-compliance, risk for being lost to follow up)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Inhibition of platelet aggregation | Pre-LD dose, 0.5, 1, 2, 3, 4-6, the next day just before and 1, 2 and 4 hours after morning maintenance dose and pre-dose and 1, 2 and 4 hours after the last study MD dose (14 +/- 3 days).
  The primary end point is the pharmacodynamic (inhibition of platelet aggregation, IPA) effect of 180mg LD ticagrelor measured at 1hour post-dose by 20uM ADP-induced maximum platelet aggregation

CONTACTS AND LOCATIONS:
Overall Officials: Paul Gurbel, MD, Principal Investigator — Sinai Center for Thrombosis Research
Locations (1):
- Sinai Center for Thrombosis Research, Baltimore, Maryland, United States